CLINICAL TRIAL: NCT03246893
Title: Efficacy of High Flow Oxygen Nasal Cannula Versus Noninvasive Positive Pressure Ventilation After Extubation in Sepsis Patients
Brief Title: Efficacy of HFNC Versus NIV for Prevent Reintubation in Sepsis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Surat Tongyoo, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Si212/2017
Record Dates: First submitted 2017-08-03; First posted 2017-08-11 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Post Extubation Respiratory Failure; Re-intubation; Septic Shock; Severe Sepsis
Keywords: Sepsis; Septic shock; Severe sepsis; Extubation; Reintubation; Noninvasive positive pressure ventilation; High flow oxygen nasal cannula
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noninvasive positive pressure ventilation (Placebo Comparator): After extubation, patient will receive non invasive positive pressure ventilation (NIV) for prevent respiratory and reintubation
  Interventions: Device: Noninvasive positive pressure ventilation
- High flow oxygen nasal cannula (Experimental): After extubation, patient will receive high flow oxygen cannula for prevent respiratory and reintubation
  Interventions: Device: High flow oxygen nasal cannula

INTERVENTIONS:
Device: Noninvasive positive pressure ventilation — Noninvasive positive pressure ventilation will apply via a face mask with initial setting as the following:
  Inspiratory pressure 6-8 cmH2O Expiratory pressure 3-5 cmH2O FiO2 30-60% Respiratory rate 12-16 per min
  Other Names: NIV
  Arms: Noninvasive positive pressure ventilation
Device: High flow oxygen nasal cannula — High flow oxygen nasal cannula will apply to patient via a nasal cannula with initial setting as the following:
  Temperature 37 degree celsius Flow 30 liter per min FiO2 40-60%
  Other Names: HFNC
  Arms: High flow oxygen nasal cannula

SUMMARY:
Post extubation respiratory failure occur in 30% of extubated patients. More than 50% of them required reintubation. Noninvasive positive pressure ventilation (NIV) had been reported as an effective tool to prevent post extubation respiratory failure. Recently, high flow oxygen nasal cannula (HFNC) had been successfully used to prevent post extubation respiratory failure and prevent reintubation in comparable with NIV among post cardiothoracic surgery and high risk for reintubated patients. There was no information about HFNC versus NIV in prevention of reintubation among severe sepsis or septic shock patients.

DETAILED DESCRIPTION:
Post extubation respiratory failure occur in 30% of extubated patients. More than 50% of them required reintubation. Noninvasive positive pressure ventilation (NIV) had been reported as an effective tool to prevent post extubation respiratory failure. Recently, high flow oxygen nasal cannula (HFNC) had been successfully used to prevent post extubation respiratory failure and prevent reintubation. The results from recent randomized controlled trials, comparing HFNC with NIV for prevent post extubation respiratory failure among post cardiac surgery and high risk patients, showed no significant different in the treatment outcome.comparable with NIV among post cardiothoracic surgery and high risk for reintubated patients.

About 40-85% of severe sepsis/septic shock patients developed acute respiratory failure, required endotracheal intubation. According to the nature of patients population, usually eldery, multiple co-morbid condition and high APACHE II score, sepsis patients were considerred as high risk for reintubation, after extubated. There was no information about HFNC versus NIV in prevention of reintubation among severe sepsis or septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sepsis or septic shock according to the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3)
* Depended on mechanical ventilator for more than 48 hours
* Plan for extubation due to successful weaning

Exclusion Criteria:

* Patient with tracheostomy
* Recent upper abdominal surgery
* Wound at face that prohibit face-mask application
* Patient or 1st degree relative not agree to participate trial
* Physician prefer either NIV or HFNC for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Device failure rate | an average of 1 year
  Device failure to prevent reintubation, patient discomfort, change to another device within 72 hours after extubation

SECONDARY OUTCOMES:
Reintubation rate | an average of 1 year
  Patient develope respiratory failure, requiring reintubation within 72 hours after extubation
28 day mortality rate | Upto 28 days
  Proportion of dead patients to overall patients
Hospital mortality rate | an average of 1 year
  Proportion of dead patients to overall patients from extubation to discharge date

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, Dr, Principal Investigator — Siriraj Hospital
Locations (1):
- Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Derived] Tongyoo S, Tantibundit P, Daorattanachai K, Viarasilpa T, Permpikul C, Udompanturak S. High-flow nasal oxygen cannula vs. noninvasive mechanical ventilation to prevent reintubation in sepsis: a randomized controlled trial. Ann Intensive Care. 2021 Sep 14;11(1):135. doi: 10.1186/s13613-021-00922-5. PMID 34523035